CLINICAL TRIAL: NCT03820557
Title: Increasing Shared Decision Making and Patient Participation in Lung Cancer Clinical Trials (Free to Breathe)
Brief Title: Decision Counseling Program in Increasing Shared Decision Making and Clinical Trial Participation in Patients With Stage 0-IV Lung Cancer (Free to Breathe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17G.352; JT 10803 (Other: JeffTrial Number)
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Counseling (Experimental): Patients undergo participation in the DCP prior to an audio-recorded oncology appointment.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Undergo Decision Counseling Program

SUMMARY:
This clinical trial studies how well the Decision Counseling Program works in increasing patient-physician shared decision making and participation in clinical trials for lung cancer patients. Decision aids help provide patients with information that may help them select a course of action related to their cancer care when more than one alternative is available. It also encourages shared decision making allowing patients and their providers to make health decisions together. Determining how patients make decisions about participating in a clinical trial may help doctors facilitate patient decision making and improve participation in lung cancer clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Facilitate patient deliberation about participation in a lung cancer clinical trial using the Decision Counseling Program (DCP).

SECONDARY OBJECTIVES:

I. Document the extent to which patient values and preferences are incorporated into physician-patient shared decision making (SDM) about cancer clinical trials.

II. Assess changes in patient knowledge, anxiety, and decisional conflict related to clinical trial participation.

III. Characterize patient and physician experience with intervention exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer (Stages 0, 1, 2, 3, 4)
* Lung cancer patients for which there is an available interventional clinical trial open at Jefferson Kimmel Cancer Center
* Patients being treated by a lung medical oncologist on the Center City Campus of Thomas Jefferson University
* Able to provide informed consent
* English-speaking

Exclusion Criteria:

* Inability to communicate in English
* Unable to provide informed consent
* Not eligible for an open, actively accruing interventional trial at Jefferson

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Patient perception related to clinical trials participation, measured by follow up survey questions | Baseline to 30 days
  Will compute descriptive statistics for all sections and determine the variables on which to compare patient responses at the two time points (baseline and endpoint) using paired t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Leader, DrPH, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/